CLINICAL TRIAL: NCT04738045
Title: Comparative Therapeutic Efficacy and Safety of Remdesivir Versus Lopinavir/ Ritonavir and Remdesivir Combination in COVID-19 Patients
Brief Title: Comparison of Remdesivir Versus Lopinavir/ Ritonavir and Remdesivir Combination in COVID-19 Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Essam (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Essam, Principle Investigator, October 6 University
Organization: October 6 University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-21001
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Remdesivir; Lopinavir/ Ritonavir
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Lopinavir; Ritonavir; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): Remdesivir will be administrated intravenously (IV) at a dose of 200 mg loading dose then 100 mg once daily for 5 days.
  Interventions: Drug: Remdesivir
- interventional (Experimental): Remdesivir will be administrated intravenously (IV) at a dose of 200 mg loading dose then 100 mg once daily and Lopinavir / ritonavir at a dose of 400 /100 once daily for 5 days.
  Interventions: Drug: Lopinavir/ Ritonavir and Remdesivir combination

INTERVENTIONS:
Drug: Remdesivir — Remdesivir will be administrated intravenously (IV) at a dose of 200 mg loading dose then 100 mg once daily.
  Other Names: control
  Arms: control
Drug: Lopinavir/ Ritonavir and Remdesivir combination — Remdesivir will be administrated intravenously (IV) at a dose of 200 mg loading dose then 100 mg once daily and Lopinavir / ritonavir at a dose of 400 /100 once daily for 5 days
  Other Names: intervention
  Arms: interventional

SUMMARY:
Comparison outcomes of a large cohort of moderate and severe COVID-19 patients received remdesivir alone with patients who received remdesivir in combination with lopinavir/ ritonavir in addition to standard management.

DETAILED DESCRIPTION:
Aim of the study

1. To assess the difference in patients' clinical status improvement between patients receiving remdesivir alone and patients receiving remdesivir and lopinavir/ ritonavir.
2. To detect time to improvement in oxygenation among both groups.
3. To detect duration of hospitalization and mortality rate in both groups.
4. To detect incidence and duration of mechanical ventilation in both treatment arms.
5. To monitor of adverse events of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients with pneumonia evidenced by chest CT scan.
* Laboratory (RT-PCR) confirmed infection with 2019-nCoV or strongly suspected to be infected with SARS-COV2 with confirmation studies pending.
* And at least one of the following:

  1. Respiratory frequency ≥30/min.
  2. Blood oxygen saturation ≤93% on room air (RA).
  3. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) <300.
  4. Worsening of lung involvement, defined as an increase in number and/or extension of pulmonary areas of consolidation, need for increased FiO2 to maintain stable O2 saturation, or worsening O2 saturation of >3% with stable FiO2.

Exclusion Criteria:

* Baseline elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 5-fold the upper limit of the normal range.
* Pregnancy.
* Known hypersensitivity to drugs or any component of the formulation.
* Serious co-morbidity, including: Hepatic patients child Pugh class C.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of cured patients in the interventional group versus the proportion of cured patients in the control group | "through study completion, an average of 3 months"
  Clinical cure will be assessed after 5-7 days from starting treatment based on:
  1. Improvement in oxygenation (SpO2/FiO2 ratio).
  2. Time to improvement in oxygenation.
  3. Duration of hospitalization.
  4. Mortality rate.

SECONDARY OUTCOMES:
Monitoring of adverse events. | "through study completion, an average of 3 months"
  The occurrence of adverse events will be recorded on a daily basis, with a focus on: bacterial or fungal infections, elevation of AST or ALT level > 3x the upper limit of normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Sarhan, PhD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef University, Banī Suwayf, Egypt